CLINICAL TRIAL: NCT00005434
Title: Opioid Compromise in Hypertension--Modulating Factors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4361; R29HL046218 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To confirm the preliminary findings of age, race, and hypertension chronicity effects on opioid and cardiovascular responses to stress and to determine the opioid mechanisms mediating these effects using an opioid receptor blockade strategy.

DETAILED DESCRIPTION:
BACKGROUND:

Opioids exert depressor effects on cardiovascular responses through sympathetic nervous system inhibition. Research suggests that opioid inhibition of sympathetic activity may be compromised in hypertension. Preliminary studies by the Principal Investigator suggest that the nature of this compromise may be influenced by age and race. Additionally, literature suggests that hypertension chronicity may modulate opioid sympathoinhibitory actions. The receptor mechanisms mediating the observed modulating effects of age, race, and hypertension chronicity on opioidergic inhibition and regulation of blood pressure remained to be determined.

DESIGN NARRATIVE:

Two double-blind, placebo-controlled cross-over studies were conducted to evaluate the effects of naltrexone hydrochloride, an oral opiate antagonist, on adrenergically-mediated cardiovascular responses in older and younger, Black and White normotensives and hypertensives with varying lengths of hypertension duration. Cardiovascular and opioid responses were measured in response to a stressor combined with either placebo or naltrexone pretreatment. Results from these studies assisted in (a) elucidating opioidergic mechanisms underlying the increased rates of hypertension morbidity and mortality among Blacks and the elderly, and (b) ultimately optimized the design of pharmacological interventions for the prevention and treatment of hypertension.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-04; Study Completion 1997-03 (Actual)

REFERENCES:
- [Background] Svetkey LP, Timmons PZ, Emovon O, Anderson NB, Preis L, Chen YT. Association of hypertension with beta2- and alpha2c10-adrenergic receptor genotype. Hypertension. 1996 Jun;27(6):1210-5. doi: 10.1161/01.hyp.27.6.1210. PMID 8641726